CLINICAL TRIAL: NCT00279981
Title: TRENDS: A Prospective Study of the Clinical Significance of Atrial Arrhythmias Detected by Implanted Device Diagnostics
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Other Study IDs: 219
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Atrial Fibrillation; Stroke; Heart Failure
Keywords: Atrial fibrillation; Stroke; Pacemaker; Implantable Cardiac Defibrillator; Resynchronization systems
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Heart Failure | interventions — Diagnosis

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: Diagnostic

SUMMARY:
The purpose of this study is to look at the heart rate and rhythm information collected daily in Medtronic implantable pulse generators (IPG), implantable cardioverter defibrillators (ICD) and cardiac resynchronization therapy (CRT) devices. The study will gather this information from many patients to see if heart rate or rhythm data can predict the risk of a patient having a medical condition such as stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent and privacy/protection authorization.
* Subjects 65 years of age or older.

OR

* Subjects with age >18 and < 65 years and one of the following stroke risk factors:
* Prior stroke or TIA
* Diagnosis of hypertension (HTN)
* Diagnosis of Diabetes Mellitus (DM)
* Diagnosis of Congestive Heart Failure (CHF)
* Subjects who meet the Class I/Class II indications for a dual chamber implantable pulse generator or dual chamber implanted cardioverter defibrillator device

OR

• Subjects who meet the criteria for indication of a dual chamber resynchronization device with bi-ventricular pacing (moderate to severe CHF symptoms [NYHA Class III-IV] despite optimal medical therapy, left ventricular ejection fraction ≤ 35%, and a QRS duration ≥130 ms)13.

Exclusion Criteria:

* Subjects who are to receive a replacement IPG, ICD or CRT device.
* Subjects with chronic (permanent) AT/AF.
* Subjects with a history of AV nodal dependent arrhythmias.
* Subjects with a terminal illness who are not expected to survive more than 6 months.
* Subjects who are unwilling or unable to cooperate or give written informed consent and privacy/protection authorization, or subjects whose legal representatives or legal guardians refuse to give informed consent or privacy/protection authorization.
* Subjects currently receiving treatment in another drug and/or device study which could affect the outcome of the trial.
* Subjects who are or will be inaccessible for follow-up at a qualified study center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3100
Dates: Start 2003-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emile Daoud, MD, Principal Investigator — Riverside Hospital; Taya Glotzer, MD, Principal Investigator — Hackensack Meridian Health
Locations (98):
- United States (92):
  - Mesa, Arizona
  - Tucson, Arizona
  - Fountain Valley, California
  - Mission Viejo, California
  - Modesto, California
  - National City, California
  - Palm Springs, California
  - Salinas, California
  - San Bernadino, California
  - Torrance, California
  - Norwalk, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Melbourne, Florida
  - Naples, Florida
  - Palm Beach Gardens, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Munster, Indiana
  - Ames, Iowa
  - Wichita, Kansas
  - Ashland, Kentucky
  - Lexington, Kentucky
  - Covington, Louisiana
  - Slidell, Louisiana
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Brighton, Massachusetts
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Grand Blanc, Michigan
  - Kalamazoo, Michigan
  - Mount Clemens, Michigan
  - Saginaw, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Gulfport, Mississippi
  - Hattiesburg, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Camden, New Jersey
  - Cherry Hill, New Jersey
  - Hackensack, New Jersey
  - Haddon Heights, New Jersey
  - West Orange, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - Greensboro, North Carolina
  - Pinehurst, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Fairview Park, Ohio
  - Marion, Ohio
  - Toledo, Ohio
  - Midwest City, Oklahoma
  - Easton, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Odessa, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - La Crosse, Wisconsin
  - Milwaukee, Wisconsin
- Australia (4):
  - Liverpool, New South Wales
  - New Lambton, New South Wales
  - Bedford Park, South Australia
  - Perth-Western Australia
- Canada (2):
  - Calgary, Alberta
  - London, Ontario

REFERENCES:
- [Derived] Yano Y, Greenland P, Lloyd-Jones DM, Daoud EG, Koehler JL, Ziegler PD. Simulation of Daily Snapshot Rhythm Monitoring to Identify Atrial Fibrillation in Continuously Monitored Patients with Stroke Risk Factors. PLoS One. 2016 Feb 16;11(2):e0148914. doi: 10.1371/journal.pone.0148914. eCollection 2016. PMID 26882334
- [Derived] Glotzer TV, Daoud EG, Wyse DG, Singer DE, Ezekowitz MD, Hilker C, Miller C, Qi D, Ziegler PD. The relationship between daily atrial tachyarrhythmia burden from implantable device diagnostics and stroke risk: the TRENDS study. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):474-80. doi: 10.1161/CIRCEP.109.849638. Epub 2009 Aug 4. PMID 19843914